CLINICAL TRIAL: NCT03441919
Title: Activation of the Innate Immune System and Vascular Inflammation in Patients With Type 1 Diabetes
Brief Title: Activation Innate Immune System in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Other Study IDs: NL62200.091.17
Record Dates: First submitted 2018-01-22; First posted 2018-02-22 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1; Cardiovascular Diseases; Innate Immune System; Inflammation; Metabolism Disorder, Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Inflammation; Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with type 1 diabetes, poor glycemic control: * Diagnosis based on clinical criteria
  * Duration of diabetes ≥10 years
  * Age ≥20 years, ≤ 60 years
  * HbA1c >64 mmol/mol
  Interventions: Radiation: PET-CT (positron emission tomography - computer tomography); Diagnostic Test: Blood drawn
- Patients with type 1 diabetes, good glycemic control: * Diagnosis based on clinical criteria
  * Duration of diabetes ≥10 years
  * Age ≥20 years, ≤ 60 years
  * HbA1c <64 mmol/mol
  Interventions: Radiation: PET-CT (positron emission tomography - computer tomography); Diagnostic Test: Blood drawn
- Healthy subjects: * Absence of disease, no use of medication
  * Matched for age, gender and BMI
  * HbA1c <42 mmol/mol
  Interventions: Radiation: PET-CT (positron emission tomography - computer tomography); Diagnostic Test: Blood drawn

INTERVENTIONS:
Radiation: PET-CT (positron emission tomography - computer tomography) — PET-CT to determine vascular inflammation
Diagnostic Test: Blood drawn — Blood drawn

SUMMARY:
Hyperglycemia is a well-known cardiovascular risk factor. It has also been shown that episodes of hyperglycemia increase the risk for cardiovascular diseases despite return to normoglycemia, a phenomenon termed 'glycemic or metabolic memory'. The molecular mechanism underlying this phenomenon remains unclear.

Cardiovascular events, such as myocardial infarction and stroke are caused by atherosclerosis, which is characterized by low grade inflammation of the vascular wall, including accumulation of innate immune cells such as monocytes and macrophages.

The investigators hypothesize that chronic hyperglycemia shifts intracellular metabolism of innate immune cells towards glycolysis and changes the epigenetic state of (progenitors of) innate immune cells (monocytes and macrophages), which reprograms these cells towards a more aggressive, pro-atherogenic phenotype, thereby accelerating atherosclerosis.

In this study, the investigators aim to test this hypothesis. This research will reveal whether the innate immune cells of patients with chronic hyperglycemia show a durable shift in intracellular metabolism and epigenetic changes and whether this associates with vascular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 and 2 (patients with type 1 diabetes):
* Diagnosis based on clinical criteria
* Duration of diabetes ≥10 years
* Age ≥20 years, ≤ 60 years
* Group 1: HbA1c >64 mmol/mol
* Group 2: HbA1c ≤64 mmol/mol
* Written informed consent

Group 3 (healthy controls):

* Absence of disease, no use of medication
* Matched for age, gender and BMI
* HbA1c <42 mmol/mol
* Written informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Smoking
* Specific Medication use:

  * Use of immunosuppressive drugs
  * Use of statins < 2 weeks before performing PET-CT (Those that use statins will be asked to discontinue for two weeks. This can be safely done in the context of primary prevention.)
  * Use of acetylsalicylic acid
* Previous cardiovascular events (ischemic stroke/TIA (transient ischemic attack), myocardial infarction, peripheral arterial disease)
* Auto-inflammatory or auto-immune diseases
* Current or recent infection (< 3 months)
* Previous vaccination (< 3 months)
* Renal failure (MDRD <45)
* BMI>30 kg/m2
* Pregnancy
* Claustrophobia
* Severe hypoglycaemia < 1 week before PET-CT

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 1 diabetes patients, without macrovascular complications. Minimum diabetes duration 10 years.
  Patients are recruited at university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Arterial wall inflammation, measured by 18F-FDG-PET/CT | through study completion, within 1 year
  Compare arterial wall inflammation (expressed as target-to-background-ratio (TBR) measured in large arterial vessels) between well- and poorly-controlled patients. The TBR is the ratio of FDG uptake in large arterial and large venous bloodvessels.

SECONDARY OUTCOMES:
FDG (fluorodeoxyglucose) uptake in spleen and bone marrow, measured by 18F-FDG-PET/CT. | through study completion, within 1 year
  Measurement of FDG uptake in bone marrow and spleen.
Inflammatory phenotype | Most measurements within 1 week after inclusion. Cytokine measurements after completion of the inclusion of all patients.
  Blood will be collected for all subjects. LPS induced TNF production
Intracellular metabolism, measured by Seahorse respirometer | within 1 day after inclusion
  Measurement of mitochondrial stress test = oxygen consumption rate (OCR)
Epigenetic changes | Within 2 months after inclusion
  Measurement of epigenetic changes by ChIP-seq (chromatin immunoprecipitation)
Arterial wall inflammation, measured by 18F-FDG-PET/CT | through study completion, within 1 year
  Compare arterial wall inflammation between diabetes patients and healthy subjects. Comparison by using TBR (see description Outcome 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Department of Internal Medicine, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thiem K, van Dierendonck XAMH, Janssen AWM, Boogaard JP, Riksen NP, Tack CJ, Stienstra R. A High Glycemic Burden Relates to Functional and Metabolic Alterations of Human Monocytes in Patients With Type 1 Diabetes. Diabetes. 2020 Dec;69(12):2735-2746. doi: 10.2337/db20-0568. Epub 2020 Sep 25. PMID 32978233